CLINICAL TRIAL: NCT02092532
Title: Open-label, Non-randomized, Unmasked, Study of IAI in Patients Which Choroidal Neovascularization Secondary to Polypoidal Choroidal Vasculopathy (PCV)
Brief Title: Intravitreal Aflibercept for Neovascular Polypoidal Choroidal Vasculopathy (RIVAL Trial)
Acronym: RIVAL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast Retina Center, Georgia (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-AMD-1401
Record Dates: First submitted 2014-03-13; First posted 2014-03-20 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Neovascular Polypoidal Choroidal Vasculopathy
MeSH Terms: interventions — 1-phenyl-3,3-dimethyltriazene; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal Aflibercept Injection (Other): All patients will receive monthly IAI 2.0 mg intravitreally for 3 months (Baseline, Months 1 and 2), followed by mandatory IAI 2.0 mg every 2 months (Months 4, 6, 8 and 10) for 12 months.
  Interventions: Drug: Rescue Intravitreal Aflibercept Injection; Procedure: Rescue Therapy with PDT, Laser or Intravitreal Steroids

INTERVENTIONS:
Drug: Rescue Intravitreal Aflibercept Injection — Patients can receive additional IAI treatment (Months 3, 5, 7, 9, and 11) if the re-treatment criteria are met.
Procedure: Rescue Therapy with PDT, Laser or Intravitreal Steroids — Starting at Month 3, patients can receive non-anti VEGF rescue therapy (ie: PDT, laser, intravitreal steroids) if the pre-defined criteria are met.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of intravitreal aflibercept injection (IAI) in patients with neovascular polypoidal choroidal vasculopathy.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, unmasked, study of IAI in patients with choroidal neovascularization secondary to polypoidal choroidal vasculopathy (PCV). Twenty treatment naïve and previously treated PCV eyes will be enrolled (only one study eye per patient will be enrolled). A maximum of 10 previously treated eyes will be enrolled. Consented, enrolled patients will be followed monthly. All patients will receive monthly IAI 2.0 mg intravitreally for 3 months (Baseline, Months 1 and 2), followed by mandatory IAI 2.0 mg every 2 months (Months 4, 6, 8 and 10) for 12 months. Patients can receive additional IAI treatment (Months 3, 5, 7, 9, and 11) if the re-treatment criteria are met. Starting at Month 3, patients can receive non-anti vascular endothelial growth factor (VEGF) rescue therapy (ie: Photodynamic Therapy (PDT), laser, intravitreal steroids) if the pre-defined criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age. Females of child bearing potential will undergo urine pregnancy testing and be required to use appropriate methods of birth control
* ICG and fluorescein angiographic characteristics consistent with active, leaking PCV with subfoveal lesions and/or subfoveal hemorrhage, lipid exudates, PED or fluid
* Best corrected early treatment of diabetic retinopathy study (ETDRS) visual acuity at 4 meters between 20/20 - 20/400 (BCVA ETDRS letter score 85 - 20 letters in the study eye)
* Lesion Characteristics - leaking lesions consistent with PCV. (No limitations on hemorrhage, fibrosis or atrophy)
* Clear ocular media to allow for photography/angiography
* Willing and able to comply with clinic visits and study-related procedures
* Patients with bilateral disease will only be able to enroll one eye
* Provide signed informed consent

Exclusion Criteria:

* Any history of systemic Anti-VEGF therapy
* Current ocular or periocular infection
* Active intraocular inflammation
* Any comorbid condition that may decrease visual acuity
* Any patients who have had intraocular surgery within the past 30 days for any condition
* For treatment naïve patients: No prior anti-VEGF, PDT, intravitreal steroids or laser (subfoveal or non foveal)
* For previously-treated patients :
* Prior anti-VEGF (ranibizumab, bevacizumab, pegaptanib) within 30 days
* Prior IAI
* Prior PDT , transpupillary thermal therapy (TTT) or radiation within 90 days (a maximum of 3 PDTs allowed)
* Prior intravitreal steroids within 90 days
* Prior non-foveal laser within 90 days
* Prior subfoveal laser
* Patients with features of dry age-related macular degeneration such as abundant drusen and symptoms/demographic features inconsistent with the diagnosis of PCV
* Allergy to fluorescein, ICG, iodine, shellfish
* Any other condition that the investigator believes would pose a significant hazard to the patient if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* History of previous subfoveal laser
* Advanced glaucoma (IOP > 25 or cup/disc ratio > 0.8)
* Pregnant or breast-feeding women
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device (IUD); bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly) *Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity | Month 6
  The primary objective of the study is the incidence and severity of ocular and systemic adverse events at Month 6.
Incidence and Severity | Month 12
  The primary objective of the study is the incidence and severity of ocular and systemic adverse events at Month 12.

SECONDARY OUTCOMES:
Change in Best Corrected Visual Acuity (BCVA) | Months 6 and 12
  •The mean change in BCVA from Baseline to Month 6 and from Baseline up to 12 months
Change in Best Corrected Visual Acuity (BCVA) | Months 6 and 12
  •Proportion of patients gaining 5, 10 and 15 letters at Months 6 and 12
Change in Best Corrected Visual Acuity (BCVA) | Months 6 and 12
  •Proportion of patients losing 5,10, and 15 letters at Months 6 and 12
Photography Assessments | Months 6 and 12
  •Mean change from baseline in central subfield thickness at Months 6 and 12 as assessed on spectral domain optical coherence tomography (SD-OCT)
Photography Assessments | Months 6 and 12
  •Mean change from baseline in macular volume at Months 6 and 12 as assessed on SD-OCT
Photography Assessments | Months 6 and 12
  •Mean change from baseline in choroidal thickness at Months 6 and 12 through SD-OCT
Photography Assessments | Months 6 and 12
  •Proportion of patients with no evidence of pigment epithelial detachment (PED), intraretinal and subretinal fluid from choroidal neovascularization (CNV) as assessed by optical coherence tomography (OCT) at 6 and 12 months
Photography Assessments | Months 6 and 12
  •Mean change from baseline in the total area of CNV fluorescein angiographic leakage at months 6 and 12
Photography Assessments | Months 6 and 12
  •Fluorescein angiograms, indocyanine green (ICG) angiograms, OCT and fundus photographs at Months 6 and 12 compared to baseline as unchanged, resolved, improved, worsened, or cannot determine. See section 9.1.2.2
Photography Assessments | Months 6 and 12
  •Rate of polyp regression and resolution at 6 and 12 Months

OTHER OUTCOMES:
Rescue Therapy | Month 12
  •Mean number of injections of IAI
Rescue Therapy | Month 12
  •Incidence of need and administration of rescue therapy with PDT, laser, or intravitreal steroids
Rescue Therapy | Month 12
  •Incidence and need of administration of additional IAI therapy

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M Marcus, MD, Principal Investigator — Part-Owner of Southeast Retina Center, PC
Locations (1):
- Southeast Retina Center, PC, Augusta, Georgia, United States